CLINICAL TRIAL: NCT02379832
Title: Pré-Eclampsie et Retard de Croissance: Une étude Longitudinale Évaluative (PERLE)
Brief Title: Pre-Eclampsia And Growth Restriction: a Longitudinal Study
Acronym: PEARL
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Chaire Jeanne-et-Jean-Louis Lévesque en périnatalogie (Unknown); Laval University (Other)
Responsible Party: Principal Investigator, Emmanuel Bujold, Principal Investigator, CHU de Quebec-Universite Laval
Other Study IDs: B14-07-2037; B14-07-2037 (Other: CER-CHU de Quebec)
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2017-07

CONDITIONS: Preeclampsia; Severe Preeclampsia; Fetal Growth Restriction; Preterm Birth
Keywords: preeclampsia; preterm birth; pregnancy; placenta; intra-uterine growth restriction; fetal growth restriction; ultrasound; doppler; biomarkers; serum; PAPP-A; PlGF; sFlt-1; endoglin
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: Samples Without DNA — Maternal serum Cord blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Nulliparous women recruited at diagnosis of preeclampsia No intervention, only observation of biochemical and ultrasonographic markers at recruitment and at delivery N= 45
- Control: Nulliparous women recruited at the beginning of pregnancy. No intervention, only observation of biochemical and ultrasonographic markers at recruitment (1st trimester), 3 other times during pregnancy (2nd and 3rd trimester) and at delivery N= 45

SUMMARY:
Preeclampsia may have several causes leading to different characteristics of the pathology. Differentiation between the "type of preeclampsia" would help to treat patients more accurately. This project aims to identify early markers that are specific to each type of preeclampsia (early or late, with or without growth restriction). Through a case-control study, many data will be collected prospectively (serum markers, ultrasonographic markers, maternal factors) among nulliparous women with no sign of preeclampsia (as soon as the first trimester) and nulliparous women with preeclampsia (at diagnosis).

DETAILED DESCRIPTION:
Background: The current definition of preeclampsia is based on signs and symptoms without reference to the pathology. The majority of preeclampsia cases would come from placental dysfunction beginning early in pregnancy, even before the onset of clinical or biochemical events leading to the diagnosis. Defects in the development of the placenta (impaired transformation of the spiral arteries) would seem to lead to poor placental perfusion. Currently, the uterine artery Doppler is the marker used to predict placental perfusion in routine monitoring of the pregnant woman. However, other placental aspects, such as the ultrasonographic measurement of placental volume could also be useful for predicting preeclampsia. Also, several studies have shown that many blood markers (PAPP-A, PlGF, sFlt-1) detected as soon as the first trimester seem effective to predict the majority of early pre-eclampsia, those occurring before 34 weeks of gestation. However, the predictive value of these markers is not so strong regarding prediction of later preeclampsia, those occurring between 34-37 weeks and at term.

Other studies show that some maternal factors, including the value of arterial pressure, BMI, maternal age, could contribute to screening for pre-eclampsia. Recent studies have also been interested in the maternal ophthalmic artery Doppler to try to predict preeclampsia even before the development of clinical symptoms.

Our hypothesis is that each of these biomarkers may be specific to a certain type of pre-eclampsia (early or late; with or without intra uterine growth restriction). We believe that actual definition of preeclampsia includes heterogenous causes and that better understanding of this pathology would help practicians to offer a more individualised treatment to their patients.

Objective: Our main goal is to characterize from a biophysical, biochemical, ultrasonographic and placental perspective the pathology of preeclampsia.

Method: This case-control study will recruit:

1. nulliparous women at 1st trimester of pregnancy. They will provide blood sample and U/S examination at 4 different times during pregnancy.
2. nulliparous women at diagnosis of preeclampsia.

Data that will be collected are:

maternal age maternal BMI maternal ethnicity maternal mean arterial pressure (at recruitment/diagnosis and delivery) gestational age at recruitment/diagnosis and at delivery maternal serum PAPP-A, PlGF, endoglin, sFlt-1 (at recruitment and delivery) cord blood PlGf, endoglin, sFlt-1 fetal crown-rump length at 1st trimester (at recruitment) fetal growth (during pregnancy) Uterine arteries Doppler Cord arteries Doppler Maternal Ophthalmic arteries Doppler Placental volume newborn birthweight

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women (no previous delivery ≥ 20 weeks)
* Expect to deliver in recruiting center
* Control group: recruited between 11 - 13 6/7 weeks of gestation
* Case group: recruited at time of diagnosis of preeclampsia > 20 weeks of gestation

Exclusion Criteria:

* multiple pregnancy
* pregnant women <18 years old at recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nulliparous pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
early onset preeclampsia | diagnosed between 20 and 34 weeks of gestation
  Preeclampsia will be defined according to the Canadian Guidelines for Diagnosis, Evaluation, and Management of the Hypertensive Disorders of Pregnancy guidelines, as de novo hypertension with diastolic blood pressure >90 mmHg on two occasions at least four hours apart, after 20 weeks of pregnancy, associated with proteinuria ≥300 mg/24 h or at least '2 +' protein on urine dipstick or an adverse conditions

SECONDARY OUTCOMES:
Fetal growth restriction | between 20 and 42 weeks of gestation
  Fetal growth restriction will be defined as a birth weight below the 10th centile (or below the 3rd centile for severe FGR) of Canadian reference growth charts.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bujold, MD, MSc, Principal Investigator — CHU de Québec
Locations (1):
- CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No